CLINICAL TRIAL: NCT02166931
Title: The Effectiveness of BRAND'S® Essence of Chicken in the Promotion of Resilience and Resistance to Stress-associated Cognitive Inhibition
Brief Title: BRAND'S® Essence of Chicken in the Promotion of Resilience and Resistance to Stress-associated Cognitive Inhibition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201306043
Record Dates: First submitted 2014-06-09; First posted 2014-06-18 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Stress Associated Cognitive Inhibition; Essence of Chicken; Cognition; Immunity; Metabolism
Keywords: Essence of Chicken; stress; cognitive function

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): placebo with the same color, order, taste as BRAND'S® Essence of Chicken , 70cc daily for 2weeks
  Interventions: Dietary Supplement: Chicken Essence
- Chicken Essence (Experimental): BRAND'S® Chicken Essence 70cc, daily for 2 weeks
  Interventions: Dietary Supplement: Chicken Essence

INTERVENTIONS:
Dietary Supplement: Chicken Essence — BRAND'S® Chicken Essence of 70cc daily for 2 weeks Placebo 70 cc daily for 2 weeks
  Other Names: BRAND'S® Chicken Essence

SUMMARY:
The purpose of this study is to determine whether BRAND'S® Essence of Chicken are effective in the promotion of resilience and resistance to stress-associated cognitive inhibition.

DETAILED DESCRIPTION:
This is a placebo-controlled, randomized, double-blind trial. There will be 100 subjects. Subjects are randomly assigned into either placebo or BRAND'S® Essence of Chicken (BEC), 70cc daily for 2 weeks, group.

Stress test, cognitive function assessment and blood tests will be carried out at Week 0, Week 2, and Week 4 (2 weeks after termination of supplementation).

The primary end-point is the better improvement of cognitive function after supplement with BEC than placebo. The second endpoints include improvement of global health survey and changes of biomarkers related to stress and immunity.

ELIGIBILITY:
Inclusion Criteria:

* aged over 20 years,
* mildly stressed with Perceive Stress Scale (PSS) score higher than 25
* All the participants should not require medication for their mood disturbance affected by stress during the trial.

Exclusion Criteria:

* history of chronic diseases
* any psychiatric or neurological diseases (e.g. depression)
* other medical illnesses (e.g. stroke, diabetes, other cardiovascular diseases)
* allergy history to chicken

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-03 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-09-18 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in cognitive function at week 2 and week 4 | baseline, week 2, week 4
  Working memory, Episodic memory, Attention

SECONDARY OUTCOMES:
Change from baseline in biomarkers and and immunity related to stress at week 2 and week 4 | baseline, week 2, week 4
  ACTH, Cortisol, Melatonin, Glucose, BUN/CRE, GOT/GPT

OTHER OUTCOMES:
Change from baseline in global health survey at week 2 and week 4 | baseline, week 2, week 4
  chinese version of SF36

CONTACTS AND LOCATIONS:
Overall Officials: Chaur-Jong Hu, M.D., Principal Investigator — Neurology, Shuang Ho Hospital, Taipei Meidcal University, New Taipei City, Taiwan
Locations (1):
- Shuang Ho Hospital, Taipei medical University, New Taipei City, Taiwan